CLINICAL TRIAL: NCT00392977
Title: Brain Manganese Deposition in High Risk Neonates
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Principal Investigator, Judy Aschner, Adjunct Professor of Pediatrics, Vanderbilt University
Other Study IDs: ES013730; ES013730
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Necrotizing Enterocolitis; Digestive System Abnormalities; Cholestasis
Keywords: Manganese; Neonatal Intensive Care; MRI; Parenteral Nutrition; Prematurity
MeSH Terms: conditions — Enterocolitis, Necrotizing; Digestive System Abnormalities; Cholestasis; Hyperphagia; Premature Birth

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Dietary Supplement: remove Mn from PN if evidence of increased brain Mn on MRI — trace element cocktail will be withheld and zinc, copper and chromium added to PN individually.

SUMMARY:
Excessive exposure to manganese (Mn) results in Mn deposition in the brain causing adverse neurological effects. Sick infants requiring parenteral nutrition (PN) may be at increased risk of Mn neurotoxicity because neonatal PN solutions contain high concentrations of Mn. This proposal will investigate brain deposition of Mn, a paramagnetic element, by magnetic resonance (MR) imaging in preterm and term neonates receiving Mn-supplemented PN and gestational age-matched control infants. The goals of this project are to identify neonatal populations that are at increased risk of excessive brain Mn deposition based on their gestational age, iron status, hepatic function and dietary Mn intake, and to make evidence-based recommendations for appropriate Mn supplementation and monitoring of infants receiving PN.

DETAILED DESCRIPTION:
Manganese (Mn) is an essential metal needed for normal growth and development. Excessive environmental or dietary exposure results in Mn deposition in Mn-sensitive brain regions causing adverse psychological and neurological effects. Sick infants requiring parenteral nutrition (PN) may be at increased risk of Mn neurotoxicity because neonatal PN solutions contain high concentrations of Mn, PN bypasses the normal intestinal absorptive control and biliary excretory mechanisms for Mn, and infants are at a critical stage of brain development. Furthermore, iron (Fe) deficiency, a common problem among sick neonates, increases Mn brain uptake because Mn and Fe compete for the same carrier transport systems in the central nervous system. This proposal will investigate brain deposition of Mn, a paramagnetic element, by magnetic resonance (MR) imaging in 40 neonates receiving Mn-supplemented PN and 10 control infants.

Two specific aims will test the following hypotheses:

1. Shortening of MR T1 and T2 relaxation times (a marker for Mn) in Mn-sensitive brain regions in neonates receiving PN will correlate directly with

   * dietary Mn intake,
   * days on PN,
   * blood Mn levels (measured by Inductively Coupled Plasma-Mass Spectrometry)
   * hepatic dysfunction/cholestasis (assessed by conjugated bilirubin levels).
2. shortening of T1 and T2 relaxation times will correlate inversely with

   * gestational age
   * Fe status (assessed by serum Fe, ferritin, transferrin, soluble transferrin receptor and hemoglobin).

The potential for increased brain Mn accumulation in infants and the potential health risks associated with elevated brain Mn burden represent crucial, unexplored issues of exposure and susceptibility. The impact of dietary Mn, and especially parenterally delivered dietary Mn, gestational age, Fe status, and hepatic dysfunction on the ability of the neonatal brain to regulate Mn deposition has not been scientifically addressed. The proposed clinical investigation has enormous health significance and may shed light on the development and progression of neurological dysfunction in infants and children on prolonged parenteral nutrition.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 30 days postnatal age
2. In the preceding four weeks have received >75% of their nutrition as Mn-supplemented PN
3. Clinically stable for transport to the MR facility
4. Signed parental consent.

Exclusion Criteria:

1. Any infant not expected to survive to the age of 3 months or
2. Not expected to achieve sufficient clinical stability to tolerate the MRI procedure.

Ages: 30 Days to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates in the NICU on prolonged PN
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2006-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Correlation between changes in MR signals and dietary Mn intake, number of days on PN and blood Mn levels | at hospital discharge and 6 months of age

SECONDARY OUTCOMES:
Comparison of pallidal-white matter T1 ratios and absolute T1 and T2 values in control infants and neonates receiving Mn-supplemented PN. | at hospital discharge and at 6 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Judy L Aschner, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt Children's Hospital, Nashville, Tennessee, United States

REFERENCES:
- [Background] Aschner JL, Aschner M. Nutritional aspects of manganese homeostasis. Mol Aspects Med. 2005 Aug-Oct;26(4-5):353-62. doi: 10.1016/j.mam.2005.07.003. PMID 16099026
- [Background] Erikson KM, Thompson K, Aschner J, Aschner M. Manganese neurotoxicity: a focus on the neonate. Pharmacol Ther. 2007 Feb;113(2):369-77. doi: 10.1016/j.pharmthera.2006.09.002. Epub 2006 Sep 22. PMID 17084903
- [Background] Fitsanakis VA, Zhang N, Avison MJ, Gore JC, Aschner JL, Aschner M. The use of magnetic resonance imaging (MRI) in the study of manganese neurotoxicity. Neurotoxicology. 2006 Sep;27(5):798-806. doi: 10.1016/j.neuro.2006.03.001. Epub 2006 Apr 18. PMID 16620989
- [Background] Fitsanakis VA, Piccola G, Marreilha dos Santos AP, Aschner JL, Aschner M. Putative proteins involved in manganese transport across the blood-brain barrier. Hum Exp Toxicol. 2007 Apr;26(4):295-302. doi: 10.1177/0960327107070496. PMID 17615110
- [Background] Yin Z, Aschner JL, dos Santos AP, Aschner M. Mitochondrial-dependent manganese neurotoxicity in rat primary astrocyte cultures. Brain Res. 2008 Apr 8;1203:1-11. doi: 10.1016/j.brainres.2008.01.079. Epub 2008 Feb 11. PMID 18313649
- [Derived] Aschner JL, Anderson A, Slaughter JC, Aschner M, Steele S, Beller A, Mouvery A, Furlong HM, Maitre NL. Neuroimaging identifies increased manganese deposition in infants receiving parenteral nutrition. Am J Clin Nutr. 2015 Dec;102(6):1482-9. doi: 10.3945/ajcn.115.116285. Epub 2015 Nov 11. PMID 26561627